CLINICAL TRIAL: NCT00096525
Title: Phase II Trial of CC-5013 in Patients With Advanced Renal Cell Carcinoma With Either No Prior Treatment or One Prior Treatment Regimen
Brief Title: Lenalidomide in Treating Patients With Advanced or Unresectable Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 04-014; MSKCC-04014
Record Dates: First submitted 2004-11-09; First posted 2004-11-10 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Lenalidomide

INTERVENTIONS:
Drug: lenalidomide

SUMMARY:
RATIONALE: Biological therapy such as lenalidomide use different ways to stimulate the immune system and stop tumor cells from growing. It may also stop the growth of tumor cells by stopping blood flow to the tumor.

PURPOSE: This phase II trial is studying how well lenalidomide works in treating patients with advanced or unresectable kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the best response in patients with advanced or unresectable renal cell cancer treated with lenalidomide (CC-5013).
* Determine the time to disease progression in patients treated with this drug.

Secondary

* Determine the safety of this drug in these patients.

OUTLINE: This is an open-label study.

Patients receive oral lenalidomide (CC-5013) once daily on days 1-21. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at 30 days and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 14-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell carcinoma (RCC)

  * Advanced or unresectable disease
* At least 1 measurable lesion
* No active brain metastases

  * Prior brain metastases allowed provided patient has been treated with radiotherapy or surgery AND remains asymptomatic for ≥ 6 months

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* No hepatitis A, B, or C infection

Renal

* Creatinine ≤ 2.0 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No known hypersensitivity to thalidomide
* No other serious medical condition, laboratory abnormality, or psychiatric illness that would preclude giving informed consent
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix or breast, localized prostate cancer, or superficial bladder cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No more than 1 prior systemic immunotherapy regimen for RCC
* No prior lenalidomide (CC-5013)
* No prior or concurrent thalidomide

Chemotherapy

* No more than 1 prior systemic chemotherapy regimen for RCC

Endocrine therapy

* No more than 1 prior systemic hormonal therapy regimen for RCC

Radiotherapy

* See Disease Characteristics
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* At least 4 weeks since prior surgery and recovered

Other

* No more than 1 other prior systemic therapy regimen for RCC
* No other concurrent anticancer therapies
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-07; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Efficacy (complete and partial response)

SECONDARY OUTCOMES:
Toxicity
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Gnanamba V. Kondagunta, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Patel PH, Kondagunta GV, Schwartz L, Ishill N, Bacik J, DeLuca J, Russo P, Motzer RJ. Phase II trial of lenalidomide in patients with metastatic renal cell carcinoma. Invest New Drugs. 2008 Jun;26(3):273-6. doi: 10.1007/s10637-007-9107-y. Epub 2007 Dec 27. PMID 18161005